CLINICAL TRIAL: NCT02647879
Title: Treatment as Prevention for Hepatitis C in Iceland. A Nationwide Campaign for Reducing Disease Burden Using Combination Antiviral Treatment
Brief Title: Treatment as Prevention for Hepatitis C in Iceland
Acronym: TraPHepC
Status: Recruiting | Type: Observational
Sponsor: Landspitali University Hospital (Other)
Collaborators: National Center of Addiction Medicine (SAA) (Other)
Responsible Party: Sponsor
Other Study IDs: LSH-15-003
Record Dates: First submitted 2015-12-30; First posted 2016-01-06 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis C infected: All patients diagnosed with hepatitis C in Iceland

SUMMARY:
The main aim of this study is to test in the Icelandic population the hypothesis that a nationwide treatment program which offers effective treatment to all known cases of Hepatitis C with the aim of halting HCV (Hepatitis C virus) transmission will lead to a reduction in incidence and disease burden associated with chronic HCV infection.

DETAILED DESCRIPTION:
In Iceland, a nationwide effort is planned where all patients with HCV infection will be offered treatment using direct acting antiviral agents. The aim of the initiative, besides offering cure to patients, is to substantially reduce domestic transmission of HCV and thereby lower the incidence. Ultimately, with these intense efforts the long-term complications of chronic HCV infection could potentially be nearly eliminated. In Iceland, there is mandatory reporting of all new cases of hepatitis C to the State Epidemiologist.

In the study, short term and long term outcomes of this initiative will be investigated. In an initial treatment phase which will last for up to three years, all patients diagnosed with hepatitis C in Iceland will be offered treatment with direct acting antiviral agents. Virological response rate and compliance will be monitored. Long term, the incidence of HCV infection acquired in Iceland will be monitored for up to 15 years, and the incidence rates of cirrhosis and hepatocellular carcinoma due to HCV will be monitored for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* HCV positive subjects 18 years and older, living in Iceland and covered by the Icelandic Health Insurance.

Exclusion Criteria:

* Age under 18 years
* Inability to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with chronic HCV infection in Iceland
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-12 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of transmission of HCV in Iceland | Measured annually for up to 15 years

SECONDARY OUTCOMES:
Incidence of cirrhosis and hepatocellular carcinoma in Iceland | Measured annually for up to 15 years
Sustained virological response rate (SVR) to treatment with antiviral agents as measured by negative HCV RNA 12 weeks post treatment | Measured for up to 36 months
Reinfection rate as measured by new infections diagnosed in patients who were previously treated and achieved SVR | Measured for up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Sigurdur Olafsson, MD, Principal Investigator — Landspitali University Hospital
Locations (1):
- Landspitali, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johannesson JM, Fridriksdottir RH, Love TJ, Runarsdottir V, Hansdottir I, Love A, Thordardottir M, Hernandez UB, Olafsson S, Gottfredsson M; Treatment as Prevention for Hepatitis C (TraP Hep C) group. High Rate of Hepatitis C Virus Reinfection Among Recently Injecting Drug Users: Results From the TraP Hep C Program-A Prospective Nationwide, Population-Based Study. Clin Infect Dis. 2022 Nov 14;75(10):1732-1739. doi: 10.1093/cid/ciac272. PMID 35438144
- [Derived] Olafsson S, Fridriksdottir RH, Love TJ, Tyrfingsson T, Runarsdottir V, Hansdottir I, Bergmann OM, Bjornsson ES, Johannsson B, Sigurdardottir B, Love A, Baldvinsdottir GE, Hernandez UB, Gudnason T, Heimisdottir M, Hellard M, Gottfredsson M. Cascade of care during the first 36 months of the treatment as prevention for hepatitis C (TraP HepC) programme in Iceland: a population-based study. Lancet Gastroenterol Hepatol. 2021 Aug;6(8):628-637. doi: 10.1016/S2468-1253(21)00137-0. Epub 2021 Jun 23. PMID 34171267
- [Derived] Olafsson S, Tyrfingsson T, Runarsdottir V, Bergmann OM, Hansdottir I, Bjornsson ES, Johannsson B, Sigurdardottir B, Fridriksdottir RH, Love A, Hellard M, Love TJ, Gudnason T, Heimisdottir M, Gottfredsson M. Treatment as Prevention for Hepatitis C (TraP Hep C) - a nationwide elimination programme in Iceland using direct-acting antiviral agents. J Intern Med. 2018 May;283(5):500-507. doi: 10.1111/joim.12740. Epub 2018 Mar 7. PMID 29512219